CLINICAL TRIAL: NCT00207571
Title: Computer-assisted STD Partner Notification
Brief Title: Partner Notification Intervention for STD Clinics.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3590; R30/CCR 019151
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Contact Tracing
Keywords: computer; video; partner notification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Computer

SUMMARY:
To help public health professionals (DIS) in interviews of patients infected with STD for the names of their sex partners, this project used a computer-based partner elicitation program before the actual DIS interview. The main outcome was the mean number of partners named by those who had the intervention versus those those who did not.

DETAILED DESCRIPTION:
The primary goal of this project is to develop and evaluate an intervention that will increase the number of people who, having been exposed to a sexual partner with chlamydia, gonorrhea or syphilis, (a) are notified and (b) receive evaluation and treatment. The intervention program will be presented entirely by an automated multimedia computer system with touch screen interface. The intervention will be tailored to user, based on demographic and recent sexual history factors. The intervention is designed to (a) motivate and prompt STD clinic clients to recall and identify sexual partners, (b) teach clinic clients a set of social skills for minimizing negative reactions while informing partners that they may be infected with an STD; (c) increase client's self-efficacy relative to disclosing partners names and informing them of their STD exposure, and (d) provide clients with tools for motivating their partners to seek treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older AND
* Anglo, Hispanic, or Black AND
* STD diagnosis positive

Exclusion Criteria:

* Non-English speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2001-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
1. Numbers of partner named.
2. Amount and quality of identifying information.

SECONDARY OUTCOMES:
1. Willingness to name partners.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hogben, PhD, Principal Investigator — Centers for Disease Control and Prevention; Christy Sherman, PhD, Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States